CLINICAL TRIAL: NCT06344949
Title: Ciprofol Versus Propofol for Tracheal Intubation in ICU Patients: a Randomized Controlled Pilot Study
Brief Title: Ciprofol Versus Propofol for Tracheal Intubation in ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2024-074
Record Dates: First submitted 2024-03-01; First posted 2024-04-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Emergency Tracheal Intubation in Critically Ill Patients
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol Group (Experimental)
  Interventions: Drug: Ciprofol
- Propofol Group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ciprofol — The sedation before tracheal intubation with Ciprofol
  Arms: Ciprofol Group
Drug: Propofol — The sedation before tracheal intubation with Propofol
  Arms: Propofol Group

SUMMARY:
The physiological reserves of critically ill patients are relatively low, and the risk of complications related to tracheal intubation in the ICU is higher than in the operating room. ICU tracheal intubation complications account for approximately 40% -45% of patients, including severe hypotension (10% -43%), severe hypoxemia (9% -25%), and cardiac arrest (2% -3%).Ciprofol is a novel 2,6-disubstituted phenol derivative that targeting γ-aminobutyric acid type A (GABAA)-receptor. There are four indications of ciprofol that have been approved by NMPA in recent two years: sedation and anesthesia in non-tracheal intubation procedure/operation, induction and maintenance of general anesthesia, sedation during intensive care, sedation and maintenance in gynecological outpatient surgery. The aim of this study is to compare the effects of propofol and propofol on the circulatory system during tracheal intubation in ICU patients, in order to provide a safer induction sedation regimen for emergency tracheal intubation in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need to undergo tracheal intubation under sedation after entering the ICU;
* Age range from 18 to 85 years old;
* Patients or their families have a full understanding of the purpose and significance of this trial, voluntarily participate in this clinical trial, and sign an informed consent form.

Exclusion Criteria:

* Patients who are allergic to the study drugs, or patients with contraindications to the study drugs;
* Patients with difficult airways (MACOCHA ≥ 3 points);
* Patients who require emergency intubation due to sudden cardiac arrest;
* Patients who require conscious intubation;
* Patients who can maintain mean arterial pressure (MAP) above 65mmHg using of one or more vasoactive drugs (equivalent (-)-noradrenaline > 0.3 μg kg min);
* In a state of imminent death;
* Pregnant and/or lactating women; Subject judged by the investigator to have any other factors unsuitable for participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
cardiovascular collapse within 30minutes from the start of the intubation procedure | 30 minutes from the the intubation procedure
  defined as occurrence of at least one of the following events: systolic blood pressure<65 mm Hg recorded at least once; systolic blood pressure<90 mm Hg for>30 minutes; SBP decreased more than 20% from baseline;new requirement for, or increase of vasopressors.

SECONDARY OUTCOMES:
Success rate of sedation | 30 minutes from the the intubation procedure
  Success rate of sedation
Successful intubation on the first attempt | 30 minutes from the the intubation procedure
  Successful intubation on the first attempt
Time from initiation of study drug administration to successful tracheal intubation (within 30 minutes) | Time from initiation of study drug administration to successful tracheal intubation (within 30 minutes)
  Time from initiation of study drug administration to successful tracheal intubation (within 30 minutes)
The incidence of cardiac arrest within 30 minutes after tracheal intubation | 30 minutes from the the intubation procedure
  The incidence of cardiac arrest within 30 minutes after tracheal intubation
The incidence of bradycardia within 30 minutes after tracheal intubation | 30 minutes from the the intubation procedure
  The incidence of bradycardia within 30 minutes after tracheal intubation
The incidence of hypoxemia within 30 minutes after tracheal intubation | 30 minutes from the the intubation procedure
  The incidence of hypoxemia within 30 minutes after tracheal intubation
new requirement or increase of vasopressors | 30 minutes from the the intubation procedure
  new requirement or increase of vasopressors
new requirement or increase of antiarrhythmic drugs | 30 minutes from the the intubation procedure
  new requirement or increase of antiarrhythmic drugs
Length of ICU stay and treatment outcome | From the start of randomization until patients were transferred out of the ICU or discharged
  Length of ICU stay and treatment outcome
28 days without mechanical ventilation | From the beginning of patients enrolled to 28 days after enrollment
  28 days without mechanical ventilation
28-day mortality rate | within 28 days
  28-day mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Admass BA, Endalew NS, Tawye HY, Melesse DY, Workie MM, Filatie TD. Evidence-based airway management protocol for a critical ill patient in medical intensive care unit: Systematic review. Ann Med Surg (Lond). 2022 Aug 4;80:104284. doi: 10.1016/j.amsu.2022.104284. eCollection 2022 Aug. PMID 36045781
- [Background] Tarwade P, Smischney NJ. Endotracheal intubation sedation in the intensive care unit. World J Crit Care Med. 2022 Jan 9;11(1):33-39. doi: 10.5492/wjccm.v11.i1.33. eCollection 2022 Jan 9. PMID 35433310
- [Background] Perbet S, De Jong A, Delmas J, Futier E, Pereira B, Jaber S, Constantin JM. Incidence of and risk factors for severe cardiovascular collapse after endotracheal intubation in the ICU: a multicenter observational study. Crit Care. 2015 Jun 18;19(1):257. doi: 10.1186/s13054-015-0975-9. PMID 26084896
- [Background] Honore PM, De Bels D, Barreto Gutierrez L, Spapen HD. Hemoadsorption therapy in the critically ill: solid base but clinical haze. Ann Intensive Care. 2019 Jan 31;9(1):22. doi: 10.1186/s13613-019-0491-1. No abstract available. PMID 30706173
- [Background] Koenig SJ, Lakticova V, Narasimhan M, Doelken P, Mayo PH. Safety of Propofol as an Induction Agent for Urgent Endotracheal Intubation in the Medical Intensive Care Unit. J Intensive Care Med. 2015 Dec;30(8):499-504. doi: 10.1177/0885066614523100. Epub 2014 Feb 17. PMID 24536033
- [Background] Luo Z, Tu H, Zhang X, Wang X, Ouyang W, Wei X, Zou X, Zhu Z, Li Y, Shangguan W, Wu H, Wang Y, Guo Q. Efficacy and Safety of HSK3486 for Anesthesia/Sedation in Patients Undergoing Fiberoptic Bronchoscopy: A Multicenter, Double-Blind, Propofol-Controlled, Randomized, Phase 3 Study. CNS Drugs. 2022 Mar;36(3):301-313. doi: 10.1007/s40263-021-00890-1. Epub 2022 Feb 14. PMID 35157236
- [Background] Wu B, Zhu W, Wang Q, Ren C, Wang L, Xie G. Efficacy and safety of ciprofol-remifentanil versus propofol-remifentanil during fiberoptic bronchoscopy: A prospective, randomized, double-blind, non-inferiority trial. Front Pharmacol. 2022 Dec 21;13:1091579. doi: 10.3389/fphar.2022.1091579. eCollection 2022. PMID 36618929
- [Background] Chen BZ, Yin XY, Jiang LH, Liu JH, Shi YY, Yuan BY. The efficacy and safety of ciprofol use for the induction of general anesthesia in patients undergoing gynecological surgery: a prospective randomized controlled study. BMC Anesthesiol. 2022 Aug 3;22(1):245. doi: 10.1186/s12871-022-01782-7. PMID 35922771
- [Background] Liang P, Dai M, Wang X, Wang D, Yang M, Lin X, Zou X, Jiang K, Li Y, Wang L, Shangguan W, Ren J, He H. Efficacy and safety of ciprofol vs. propofol for the induction and maintenance of general anaesthesia: A multicentre, single-blind, randomised, parallel-group, phase 3 clinical trial. Eur J Anaesthesiol. 2023 Jun 1;40(6):399-406. doi: 10.1097/EJA.0000000000001799. Epub 2023 Jan 19. PMID 36647565